CLINICAL TRIAL: NCT05740072
Title: Effect of Drying Before Plastic Wrapping on Thermal Losses in Very Preterm Infants at Birth: a Multicenter, Randomized Controlled Trial
Brief Title: Effect of Drying Before Plastic Wrapping on Thermal Losses in Very Preterm Infants at Birth
Acronym: NEODRY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Associate Professor, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEOUNIPD2(2023)
Record Dates: First submitted 2023-02-07; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Temperature Regulation; Disorder, Fetus or Newborn
Keywords: Newborn; Prematurity; Temperature; Delivery
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drying before wrapping (Experimental): Immediately after birth, the infant's body will be dried before wrapping in a plastic bag
  Interventions: Other: Drying before wrapping
- No drying before wrapping (Active Comparator): Immediately after birth, the infant will be wrapped in a plastic bag without drying
  Interventions: Other: No drying before wrapping

INTERVENTIONS:
Other: Drying before wrapping — Immediately after birth, the infant's body will be dried before wrapping in a plastic bag
  Arms: Drying before wrapping
Other: No drying before wrapping — Immediately after birth, the infant will be put in a plastic bag without wrapping
  Arms: No drying before wrapping

SUMMARY:
This is a multicenter, unblinded, randomized controlled trial comparing drying vs. not drying before plastic wrapping for the thermoregulation of very preterm infants at birth. The aim of this study will be to compare two modes of thermal management (plastic wrapping with or without drying) for preventing heat loss at birth in very preterm infants.

DETAILED DESCRIPTION:
Background: Hypothermia in preterm infants during the immediate postnatal phase is associated with morbidity and mortality and remains an unresolved, worldwide challenge.

A list of interventions, including adequate room temperature, use of infant warmers, polyethylene bags/wrap, pre-heated mattresses, caps and heated and humidified gases, to prevent thermal loss at birth in very preterm infants has been recommended, but a certain percentage of very preterm infants are hypothermic at the time of the neonatal intensive care unit (NICU) admission suggesting that further measures are needed. While drying is recommended for the thermal management of infants with gestational age >32 weeks, this procedure is not indicated for very preterm infants who should be put in a plastic wrap immediately at birth without drying. However, such indication is based on studies comparing wrapping without drying vs. drying without wrapping, while the potential advantages of combining these interventions were not explored. We hypothesized that drying before wrapping could prevent heat loss immediately after birth and reduce hypothermia at NICU admission in very preterm infants.

Objective: The aim of this study will be to compare two modes of thermal management (plastic wrapping with or without drying) for preventing heat loss at birth in very preterm infants.

Methods: This is a multicenter, unblinded, randomized controlled trial comparing drying vs. not drying before plastic wrapping for the thermoregulation of very preterm infants at birth. After obtaining parental consent, all infants with estimated birth weight <1500 g and/or gestational age ≤30+6 weeks will be assigned to be managed with or without drying before plastic wrapping. Room temperature and maternal temperature will be measured at the time of delivery. Patients allocated in both groups will be managed based on the current guidelines for neonatal resuscitation. The primary outcome measure will be the proportion of neonates in the normal thermal range (temperature 36.5-37.5°C) at NICU admission. Secondary outcome measures will be: proportion of neonates with hypothermia (<36.5°C and <36.0°C) at NICU admission; proportion of hyperthermic neonates (temperature >37.5°C) at NICU admission; temperature at 1 hour after NICU admission; proportion of intraventricular hemorrhage; proportion of respiratory distress syndrome; proportion of late onset sepsis; proportion of bronchopulmonary dysplasia; mortality before hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Estimated birth weight <1500 g and/or gestational age ≤30+6 weeks (and)
* Inborn (and)
* Parental consent; written informed consent will be obtained by a member of the neonatal team involved in the study from a parent or guardian at the maternal admission to the Obstetric Department.

Exclusion Criteria:

* Major congenital malformations (i.e. cardiac disease, defects of abdominal wall, ...);
* Outborn;
* Parental refusal to participate in the study.

Ages: 0 Minutes to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 346 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Number (percentage) of neonates in the normal thermal range (temperature 36.5-37.5°C) at Neonatal Intensive Care Unit admission. | 25 minutes

SECONDARY OUTCOMES:
Number (percentage) of neonates with hypothermia (temperature <36.5°C) at neonatal intensive care unit admission | 25 minutes
Number (percentage) of neonates with moderate-severe hypothermia (temperature <36.0°C) at neonatal intensive care unit admission | 25 minutes
Number (percentage) of neonates hyperthermia (temperature >37.5°C) at NICU admission at neonatal intensive care unit admission | 25 minutes
Temperature at 1 hour after neonatal intensive care unit admission | 60 minutes
  Axillary temperature will be registered at 1 hour after neonatal intensive care unit admission
Number (percentage) of infants with intraventricular hemorrhage (all grades and grade III-IV) | 10 days
  The grade of intraventricular hemorrhage will be defined on Levine classification
Number (percentage) of infants with respiratory distress syndrome | 72 hours
  Respiratory distress syndrome will be defined as presence of clinical signs of respiratory distress and radiological findings
Number (percentage) of infants with late-onset sepsis | 7 days
  Sespsis will be defined based on the presence of a positive blood colture 72 hours after birth
Number (percentage) of infants with bronchopulmonary dysplasia | 36 postnatal weeks
  Bronchopulmonary dysplasia will be defined as the need for oxygen at 36 postnatal weeks gestation
Number (percentage) of infants died before hospital discharge | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers upon motivated request

REFERENCES:
- [Background] Lunze K, Bloom DE, Jamison DT, Hamer DH. The global burden of neonatal hypothermia: systematic review of a major challenge for newborn survival. BMC Med. 2013 Jan 31;11:24. doi: 10.1186/1741-7015-11-24. PMID 23369256
- [Background] Wyckoff MH, Wyllie J, Aziz K, de Almeida MF, Fabres JW, Fawke J, Guinsburg R, Hosono S, Isayama T, Kapadia VS, Kim HS, Liley HG, McKinlay CJD, Mildenhall L, Perlman JM, Rabi Y, Roehr CC, Schmolzer GM, Szyld E, Trevisanuto D, Velaphi S, Weiner GM; Neonatal Life Support Collaborators. Neonatal Life Support 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Resuscitation. 2020 Nov;156:A156-A187. doi: 10.1016/j.resuscitation.2020.09.015. Epub 2020 Oct 21. PMID 33098917
- [Background] Madar J, Roehr CC, Ainsworth S, Ersdal H, Morley C, Rudiger M, Skare C, Szczapa T, Te Pas A, Trevisanuto D, Urlesberger B, Wilkinson D, Wyllie JP. European Resuscitation Council Guidelines 2021: Newborn resuscitation and support of transition of infants at birth. Resuscitation. 2021 Apr;161:291-326. doi: 10.1016/j.resuscitation.2021.02.014. Epub 2021 Mar 24. PMID 33773829
- [Background] Trevisanuto D, Testoni D, de Almeida MFB. Maintaining normothermia: Why and how? Semin Fetal Neonatal Med. 2018 Oct;23(5):333-339. doi: 10.1016/j.siny.2018.03.009. Epub 2018 Mar 21. PMID 29599071
- [Background] Cavallin F, Doglioni N, Allodi A, Battajon N, Vedovato S, Capasso L, Gitto E, Laforgia N, Paviotti G, Capretti MG, Gizzi C, Villani PE, Biban P, Pratesi S, Lista G, Ciralli F, Soffiati M, Staffler A, Baraldi E, Trevisanuto D; Servo COntrol for PReterm Infants (SCOPRI) Trial Group. Thermal management with and without servo-controlled system in preterm infants immediately after birth: a multicentre, randomised controlled study. Arch Dis Child Fetal Neonatal Ed. 2021 Nov;106(6):572-577. doi: 10.1136/archdischild-2020-320567. Epub 2021 Feb 17. PMID 33597230